CLINICAL TRIAL: NCT00000892
Title: Activity of the Soft Gelatin Capsule of Saquinavir (SQVsgc) in Combination With Ritonavir or Nelfinavir and Combinations of Delavirdine and/or Adefovir Dipivoxil in HIV-Infected Subjects With Prior Indinavir Use and Viral Loads From 2,000 to 200,000 Copies HIV RNA/ml
Brief Title: A Study of Several Anti-HIV Drug Combinations in HIV-Infected Patients Who Have Used Indinavir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 359; 11324 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Indinavir; RNA, Viral; Saquinavir; Delavirdine; Nelfinavir; Adenine; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Carnitine; adefovir dipivoxil; Saquinavir; Delavirdine

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Levocarnitine
Drug: Adefovir dipivoxil
Drug: Saquinavir
Drug: Delavirdine mesylate

SUMMARY:
To compare the proportion of patients whose plasma HIV-1 RNA is below 500 copies/ml after 16 weeks of treatment. To assess the safety, toxicity, and tolerance of each treatment arm.

While indinavir is currently the most commonly prescribed protease inhibitor, the optimal therapy for a person on an indinavir-containing regimen who experiences a rebound in viral load or never experiences a decrease in viral load below 500 copies per milliliter is unknown. Current clinical practice for such patients typically involves empiric use of a combination of other protease inhibitors (saquinavir/nelfinavir or saquinavir/ritonavir) and at least 1 other antiretroviral agent to which the patient has had little or no prior exposure. This may involve the use of 1 or more reverse transcriptase inhibitors (RTIs) or nonnucleoside reverse transcriptase inhibitors (NNRTIs). This study attempts to formally evaluate some of these options in indinavir-experienced patients.

DETAILED DESCRIPTION:
While indinavir is currently the most commonly prescribed protease inhibitor, the optimal therapy for a person on an indinavir-containing regimen who experiences a rebound in viral load or never experiences a decrease in viral load below 500 copies per milliliter is unknown. Current clinical practice for such patients typically involves empiric use of a combination of other protease inhibitors (saquinavir/nelfinavir or saquinavir/ritonavir) and at least 1 other antiretroviral agent to which the patient has had little or no prior exposure. This may involve the use of 1 or more reverse transcriptase inhibitors (RTIs) or nonnucleoside reverse transcriptase inhibitors (NNRTIs). This study attempts to formally evaluate some of these options in indinavir-experienced patients.

Patients are stratified by HIV RNA (2,000 - 20,000 copies/ml versus 20,000 - 200,000 copies/ml), and randomized to 1 of 6 treatment arms as follows:

Arm A: Saquinavir (SQV) plus ritonavir (RTV) plus delavirdine (DLV) plus adefovir dipivoxil placebo.

Arm B: SQV plus RTV plus DLV placebo plus adefovir dipivoxil. Arm C: SQV plus RTV plus DLV plus adefovir dipivoxil. Arm D: SQV plus nelfinavir (NFV) plus DLV plus adefovir dipivoxil placebo. Arm E: SQV plus NFV plus DLV placebo plus adefovir dipivoxil. Arm F: SQV plus NFV plus DLV plus adefovir dipivoxil. In addition to assigned study treatment patients receive an L-carnitine supplement.

Therapy is administered for 24 weeks. Patients who have an average HIV RNA value for Weeks 12 and 16 that is less than 5,000 copies or a least 1 log below their baseline value may continue their assigned study treatment for an additional 24 weeks. [AS PER AMENDMENT 3/30/98: Subjects with plasma HIV RNA greater than 5,000 copies/ml may elect to continue or discontinue study medications in the treatment extension and seek the best available treatment.] [AS PER AMENDMENT 06/11/98: The dose of adefovir dipivoxil is reduced at or after Week 16. Alternatively, patients may discontinue adefovir dipivoxil/placebo and substitute appropriate antiretroviral agent(s) or add appropriate antiretroviral agent(s) to their reduced-dose regimen. Also, at the discretion of the protocol chairperson, patients who have been on study for more than 16 weeks may substitute appropriate FDA-approved antiretroviral agent(s) for any study medication that must be discontinued because of toxicity. Addition of nonnucleoside reverse transcriptase inhibitors, protease inhibitors, or investigational agents is specifically excluded.]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Chemoprophylaxis for Pneumocystis carinii pneumonia for all patients who have a CD4 cell count of equal or less than 200 cells/mm3.

Allowed:

* Topical and oral antifungal agents except ketoconazole and itraconazole.
* Treatment, maintenance or chemoprophylaxis with approved agents for opportunistic infections.
* Antibiotics.
* Systemic corticosteroids for 21 days or less for acute problems.
* Recombinant erythropoietin (rEPO) and granulocyte-colony stimulating factor (G-CSF, filgrastim).
* Regularly prescribed medications such as antipyretics, analgesics, allergy medications, antidepressants, sleep medications, oral contraceptives (not as a sole form of birth control), megestrol acetate, or testosterone.
* Alternative therapies, such as vitamins, acupuncture, and visualization techniques.
* [AS PER AMENDMENT 3/30/98: Calcium channel blockers may be used only with caution.]

Patients must have:

* HIV-1 infection documented by a licensed ELISA and confirmed by Western blot, HIV culture, HIV antigen, plasma HIV RNA, or a second antibody test other than ELISA.
* 2,000 to 200,000 HIV-1 RNA copies/ml as measured by any Roche-certified laboratory [AS

PER AMENDMENT 3/30/98:

* using the Roche Amplicor HIV-1 Monitor] within 30 days of study entry.
* Signed, informed consent from parent or legal guardian for patients less than 18 years of age.

Prior Medication: Required:

* More than 6 months cumulative indinavir therapy.
* Stable indinavir-containing antiretroviral regimen for at least 4 weeks [2 weeks AS PER AMENDMENT 3/30/98] prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Any active infection requiring acute treatment within 30 days [21 days AS PER AMENDMENT 3/30/98] prior to study entry.
* Unexplained temperature greater than 38.5 degrees for any 7 consecutive days within 30 days prior to study entry.
* Malignancy, including Kaposi's sarcoma, that requires systemic chemotherapy.

Concurrent Medication:

Excluded:

* Non-protocol-specified immunomodulatory and/or antiretroviral agents.
* Systemic cytotoxic chemotherapy.
* Ketoconazole, itraconazole, rifampin, rifabutin, alprazolam, amiodarone, astemizole, bepridil, bupropion, cisapride, clorazepate, clozapine, diazepam, encainide, estazolam, flecainide, flurazepam, isotretinoin, meperidine, midazolam, piroxicam, propafenone, propoxyphene, quinidine, terfenadine, triazolam, zolpidem, phenytoin, phenobarbital, carbamazepine, and ergot alkaloids and [ AS PER AMENDMENT 3/30/98: dexamethasone, ergot derivatives, and pimozide].

Avoided:

* Herbal medications.

Prior Medication:

Excluded:

* At least 2 weeks or more total ritonavir and/or saquinavir (hard gelatin capsule).
* NNRTIs (nevirapine, delavirdine, DMP-266, etc.), saquinavir (soft gelatin capsule), nelfinavir, 141W94VX-478, and adefovir dipivoxil.
* Immunomodulator [systemic immunomodulator AS PER AMENDMENT 3/30/98] or investigational drug therapy within 30 days prior to entry.
* Active immunization within 30 days [21 days AS PER AMENDMENT 3/30/98] prior to entry.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Study Completion 1999-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Gulick, Study Chair; D Katzenstein, Study Chair
Locations (45):
- United States (45):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - St Vincent's Hosp / Mem Sloan-Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Med Ctr, Pittsburgh, Pennsylvania
  - Brown Univ School of Medicine, Providence, Rhode Island
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Gulick RM, Hu XJ, Fiscus S, Fletcher CV, Haubrich R, Cheng H, Lagakos S, Acosta E, Swanstrom R, Mills C, Snyder S, Fischl M, Pettinelli C, Katzenstein D. Durability of salvage therapy with saquinavir SGC (SQV) in combination with ritonavir (RTV) or nelfinavir (NFV) plus delavirdine (DLV), adefovir dipivoxil (ADV), or both; ACTG 359: 48-week final results. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 338)
- [Background] Acosta EP, Gulick R, Katzenstein D, Haubrich R, Fischl M, Raasch R, Mills C, Pettinelli C, Remmel RP, Fletcher CV. Pharmacokinetic (PK) evaluation of saquinavir soft gel capsules (SQV)/ritonavir (RTV) or sqv/nelfinavir (NFV) in combination with delavirdine (DLV) and/or adefovir dipivoxil (ADV) - - ACTG 359. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:136 (abstract no 365)
- [Background] Gulick RM, et al. Salvage therapy with saquinavir sgc (SQV) in combination with ritonavir (RTV) or nelfinavir (NFV) and delavirdine (DLV), adefovir dipivoxil (ADV), or both-ACTG 359. Second International Workshop on Salvage Therapy for HIV Infection. 1999 May 19-21
- [Background] Fletcher CV, Testa MA, Haubrich R, Brundage R, Jiang H, Ickovics J, Martinez A, Snyder S, Gulick R. Relationships among Four Measures of Medication Adherence and Virologic Response in ACTG 359. 10th Conference on Retroviruses and Oppurtunistic Infections. Feb 2003. Abstract 577.
- [Result] Gulick RM, Hu XJ, Fiscus SA, Fletcher CV, Haubrich R, Cheng H, Acosta E, Lagakos SW, Swanstrom R, Freimuth W, Snyder S, Mills C, Fischl M, Pettinelli C, Katzenstein D. Randomized study of saquinavir with ritonavir or nelfinavir together with delavirdine, adefovir, or both in human immunodeficiency virus-infected adults with virologic failure on indinavir: AIDS Clinical Trials Group Study 359. J Infect Dis. 2000 Nov;182(5):1375-84. doi: 10.1086/315867. Epub 2000 Oct 9. PMID 11023461
- [Result] Gulick RM, Hu XJ, Fiscus SA, Fletcher CV, Haubrich R, Cheng H, Acosta E, Lagakos SW, Swanstrom R, Freimuth W, Snyder S, Mills C, Fischl M, Pettinelli C, Katzenstein D. Durability of response to treatment among antiretroviral-experienced subjects: 48-week results from AIDS Clinical Trials Group Protocol 359. J Infect Dis. 2002 Sep 1;186(5):626-33. doi: 10.1086/342681. Epub 2002 Aug 9. PMID 12195349
- [Result] Fletcher CV, Jiang H, Brundage RC, Acosta EP, Haubrich R, Katzenstein D, Gulick RM. Sex-based differences in saquinavir pharmacology and virologic response in AIDS Clinical Trials Group Study 359. J Infect Dis. 2004 Apr 1;189(7):1176-84. doi: 10.1086/382754. Epub 2004 Mar 16. PMID 15031785
- [Result] Swanstrom R, Bosch RJ, Katzenstein D, Cheng H, Jiang H, Hellmann N, Haubrich R, Fiscus SA, Fletcher CV, Acosta EP, Gulick RM; AIDS Clinical Trials Group Protocol 359 Team. Weighted phenotypic susceptibility scores are predictive of the HIV-1 RNA response in protease inhibitor-experienced HIV-1-infected subjects. J Infect Dis. 2004 Sep 1;190(5):886-93. doi: 10.1086/422692. Epub 2004 Jul 23. PMID 15295692
- [Result] Fletcher CV, Testa MA, Brundage RC, Chesney MA, Haubrich R, Acosta EP, Martinez A, Jiang H, Gulick RM. Four measures of antiretroviral medication adherence and virologic response in AIDS clinical trials group study 359. J Acquir Immune Defic Syndr. 2005 Nov 1;40(3):301-6. doi: 10.1097/01.qai.0000180078.53321.6a. PMID 16249704
- [Result] Haubrich RH, Jiang H, Swanstrom R, Bates M, Katzenstein D, Petch L, Fletcher CV, Fiscus SA, Gulick RM; AIDS Clinical Trials Group Protocol 359 Team. Non-nucleoside phenotypic hypersusceptibility cut-point determination from ACTG 359. HIV Clin Trials. 2007 Mar-Apr;8(2):63-7. doi: 10.1310/hct0802-63. PMID 17507321